CLINICAL TRIAL: NCT03195023
Title: Effect of Renin-angiotensin-system (RAS) Blocker Drugs on Chronic Kidney Disease (CKD) Progression in Elderly Patients With Non Proteinuric Nephropathies (PROERCAN01)
Brief Title: Effect of RAS Blockers on CKD Progression in Elderly Patients With Non Proteinuric Nephropathies (PROERCAN01)
Acronym: PROERCAN01
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Maria Maria Angeles Goicoechea Diezhandino, Nefrologist, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROERCAN01
Record Dates: First submitted 2017-06-14; First posted 2017-06-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Renal Insufficiency, Chronic; Proteinuria
Keywords: Renal insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Lisinopril; Angiotensin-Converting Enzyme Inhibitors; Amlodipine; lercanidipine; Furosemide; Thiazides

ARMS (2):
- RAS Blockers (Active Comparator): Patients in this arm will receive Lisinopril 20mg/day
  Interventions: Drug: Lisinopril
- Non RAS Blockers (Active Comparator): Patients in this arm will receive Amlodipine 10mg/day or Lercanidipine 20mg/day +/- diuretics
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Lisinopril
  Other Names: Angiotensin converting enzyme inhibitors
  Arms: RAS Blockers
Drug: Amlodipine — Patients in this arm will receive antihypertensive treatment different from RAS blockers. If they previously received RAS blockers, they will be substitute for either Amlodipine or Lercanidipine +/- diuretics
  Other Names: Lercanidipine, Furosemide, Thiazides
  Arms: Non RAS Blockers

SUMMARY:
This study evaluates the effect of renin-angiotensin blockers on chronic kidney disease progression in elderly (>65 years old) patients with non-proteinuric nephropathies. Half of the patients will receive angiotensin converting enzyme inhibitors, while the other half will not receive them. Renal function, proteinuria and cardiovascular events will be follow up during a three year period.

DETAILED DESCRIPTION:
STUDY DESIGN: Open, multicentre, prospective, parallel-group, randomized controlled study comparing the effect of an angiotensin converting enzyme inhibitor (ACEI) vs standard antihypertensive treatment without ACEI, in the progression of renal disease in elderly patients with non-proteinuric 3-4 stage chronic renal disease.

Elderly patients (> 65 years) with moderate-severe non-proteinuric chronic renal disease (estimated Glomerular Filtrate Rate between 19-59 ml per minute per 1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration Group equation) and urine-creatinine rate < 30 mg/g, will be included. They will be randomly assigned in a 1:1 ratio to receive ACEI or standard antihypertensive treatment. Patients will be followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years
* Chronic kidney disease stage 3 or 4 (GFR measured by CKD-EPI 15-59 ml/min/1,73 m2)
* Albumine/creatinine index < 30 mg/g in simple urine sample or albuminuria < 30 mg/day in 24-hour urine sample.
* Previous hypertensive treatment::

  1. patients who have not received RAS blockers in the three months prior to inclusion can be included
  2. patients who are receiving RAS blockers could be included after one month washout period

Exclusion Criteria:

* Diabetes mellitus (type 1 or 2)
* Glomerulopathy
* Chronic heart failure or coronary heart disease
* Poorly controlled hypertension (>160/100 mmHg)
* Monorrenal
* Active malignant neoplasia (except skin cancer different from melanoma). Patients who have been free of malignancy for the last 5 years could be included.
* Chronic symptomatic or not controlled inflammatory disease (eg rheumatoid arthritis, Chron disease, ulcerative colitis or systemic lupus erythematosus)
* Chronic liver disease
* Allergy or intolerance to renin angiotensin system blockers or calcium channel blockers
* Hepatitis B, C or HIV infection
* Immunosuppressive treatment in the 3 months prior to inclusion
* Hospitalization of any cause in the three months prior to inclusion
* Rapidly progressive kidney disease (decline in GFR >5ml/min/1.73 m2/year)
* Inability to sign the informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Chronic kidney disease progression | 3 years
  Increase of baseline creatinine during follow up period

SECONDARY OUTCOMES:
Security of RAS blockers in elderly patients | 3 years
  Evaluate the frequency of hiperpotassemia (K>5.5 mmol/l)
Security of RAS blockers in elderly patients | 3 years
  Evaluate the frequency of acute kidney failure (>Cr 0.3 mg/dl)
Effect of RAS blockers on mortality in elderly patients | 3 years
  Evaluate the number and cause of deaths in the study population
Effects of RAS blockers on cardiovascular risk in elderly patients | 3 years
  Evaluate and classify cardiovascular events (heart failure, acute coronary syndrome, peripheral vasculopathy) during the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Maria Angeles Goicoechea, PhD, MD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Gregorio Maranon Hospital, Madrid, Spain

REFERENCES:
- [Background] Jafar TH, Stark PC, Schmid CH, Landa M, Maschio G, de Jong PE, de Zeeuw D, Shahinfar S, Toto R, Levey AS; AIPRD Study Group. Progression of chronic kidney disease: the role of blood pressure control, proteinuria, and angiotensin-converting enzyme inhibition: a patient-level meta-analysis. Ann Intern Med. 2003 Aug 19;139(4):244-52. doi: 10.7326/0003-4819-139-4-200308190-00006. PMID 12965979
- [Background] Wright JT Jr, Bakris G, Greene T, Agodoa LY, Appel LJ, Charleston J, Cheek D, Douglas-Baltimore JG, Gassman J, Glassock R, Hebert L, Jamerson K, Lewis J, Phillips RA, Toto RD, Middleton JP, Rostand SG; African American Study of Kidney Disease and Hypertension Study Group. Effect of blood pressure lowering and antihypertensive drug class on progression of hypertensive kidney disease: results from the AASK trial. JAMA. 2002 Nov 20;288(19):2421-31. doi: 10.1001/jama.288.19.2421. PMID 12435255
- [Background] O'Hare AM, Kaufman JS, Covinsky KE, Landefeld CS, McFarland LV, Larson EB. Current guidelines for using angiotensin-converting enzyme inhibitors and angiotensin II-receptor antagonists in chronic kidney disease: is the evidence base relevant to older adults? Ann Intern Med. 2009 May 19;150(10):717-24. doi: 10.7326/0003-4819-150-10-200905190-00010. PMID 19451579
- [Background] Ahmed AK, Kamath NS, El Kossi M, El Nahas AM. The impact of stopping inhibitors of the renin-angiotensin system in patients with advanced chronic kidney disease. Nephrol Dial Transplant. 2010 Dec;25(12):3977-82. doi: 10.1093/ndt/gfp511. Epub 2009 Oct 10. PMID 19820248
- [Background] Weiss JW, Thorp ML, O'Hare AM. Renin-angiotensin system blockade in older adults with chronic kidney disease: a review of the literature. Curr Opin Nephrol Hypertens. 2010 Sep;19(5):413-9. doi: 10.1097/MNH.0b013e32833b8d6b. PMID 20539228
- [Background] Turgut F, Balogun RA, Abdel-Rahman EM. Renin-angiotensin-aldosterone system blockade effects on the kidney in the elderly: benefits and limitations. Clin J Am Soc Nephrol. 2010 Jul;5(7):1330-9. doi: 10.2215/CJN.08611209. Epub 2010 May 24. PMID 20498247
- [Derived] Garcia-Prieto AM, Verdalles U, de Jose AP, Arroyo D, Aragoncillo I, Barbieri D, Camacho RE, Goicoechea M. Renin-angiotensin-aldosterone system blockers effect in chronic kidney disease progression in hypertensive elderly patients without proteinuria: PROERCAN trial. Hipertens Riesgo Vasc. 2024 Apr-Jun;41(2):95-103. doi: 10.1016/j.hipert.2023.11.005. Epub 2024 Mar 19. PMID 38508877